CLINICAL TRIAL: NCT07088757
Title: Low-Dose Versus Standard-Dose Rectal Indomethacin to Prevent Post-Endoscopic Retrograde Cholangiopancreatography Pancreatitis: A Multicentre, Non-Inferiority, Double-Blind, Randomised, Controlled Trial
Brief Title: Low-Dose vs Standard-Dose Indomethacin for Preventing Post-ERCP Pancreatitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Ruijin Hospital (Other); Shanghai General Hospital, China (Other); Jinhua Central Hospital (Other); Taizhou Enze Medical Center Group (Other); Dongyang People's Hospital (Other); Shaoxing People's Hospital (Other); First Affiliated Hospital of Ningbo University (Network); Affiliated Hospital of Jiaxing University (Other); People's Hospital of Quzhou (Other); Zhuji People's Hospital of Zhejiang Province (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INSPIRE
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Post-ERCP Pancreatitis
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low dose indomethacin (Experimental): patients randomized to this intervention receive 50mg indomethacin
  Interventions: Drug: low dose indomethacin
- standard dose indomethacin (Active Comparator): patients randomized to this intervention receive 100mg indomethacin
  Interventions: Drug: standard dose indomethacin

INTERVENTIONS:
Drug: standard dose indomethacin — Patients randomized to this intervention receive 100mg indomethacin suppositories within 30 min before ERCP.
  Arms: standard dose indomethacin
Drug: low dose indomethacin — Patients randomized to this intervention receive 50mg indomethacin suppositories within 30 min before ERCP.
  Arms: low dose indomethacin

SUMMARY:
Endoscopic Retrograde Cholangiopancreatography (ERCP) is a widely used procedure for diagnosing and treating pancreatic and biliary diseases. Despite its benefits, ERCP carries a risk of post-procedure pancreatitis (PEP), which occurs in approximately 12.2% of cases and can significantly increase healthcare costs and patient morbidity. Preventing PEP is crucial for improving patient outcomes and reducing the economic burden of ERCP.

Nonsteroidal anti-inflammatory drugs (NSAIDs), such as indomethacin, have been shown to be effective in reducing the incidence of PEP when administered rectally before ERCP. The standard dose recommended by guidelines is 100mg, which has been associated with a significant reduction in PEP rates. However, higher doses of NSAIDs can increase the risk of adverse events, including gastrointestinal bleeding and renal impairment. Therefore, there is a need to determine whether a lower dose can provide similar benefits without increasing these risks.

This multicenter, non-inferiority, double-blind, randomized controlled trial will be conducted in China. Participants will be adults aged 18 or older scheduled for ERCP. They will be randomly assigned in a 1:1 ratio to either the low-dose (50mg) or standard-dose (100mg) indomethacin group. The intervention will be administered rectally 30 minutes before the ERCP procedure. The study will follow a double-blind design, ensuring that both patients and investigators are unaware of the treatment allocation.

The results of this trial could significantly influence clinical practice by providing evidence on the effectiveness of a lower dose of indomethacin in preventing PEP. This could lead to a reduction in the risk of adverse events associated with higher doses and potentially decrease healthcare costs without compromising patient safety. By optimizing the dosing of indomethacin, this study aims to improve the safety and cost-effectiveness of ERCP procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Patients planned to undergo Endoscopic Retrograde Cholangiopancreatography

Exclusion Criteria:

* Standard contraindications to ERCP
* Allergy to Nonsteroidal Anti-Inflammatory Drugs (NSAIDs)
* Use of NSAIDs within 7 days prior to ERCP
* Not suitable for NSAIDs administration (gastrointestinal hemorrhage within 4 weeks, renal dysfunction [Cr >1.4mg/dl=120umol/l]; presence of coagulopathy before the procedure)
* Acute pancreatitis within 3 days before ERCP
* Hemodynamic instability
* Pregnancy or lactation
* Patients who are unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1366 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The Proportion of Subjects in Each Study Group With Post-ERCP Pancreatitis | Within 48 hours after ERCP

SECONDARY OUTCOMES:
The Proportion of Subjects in Each Study Group With Moderate-severe Post-ERCP Pancreatitis | Within one month of ERCP
Rate of Overall ERCP-related complications | Within one month of ERCP
  ERCP-related complications include post-ERCP pancreatitis, gastrointestinal bleeding, perforation or infection according to Cotton Criteria.
Rate of ERCP-related perforation | Within one month of ERCP
Rate of ERCP-related infection | Within one month of ERCP
Rate of ERCP-related bleeding | Within one month of ERCP
Rate of NSAIDs-related complications | Within one month of ERCP
  NSAIDs-related complications include: acute kidney injury, allergic reaction, gastrointestinal bleeding, myocardial infarction, cerebrovascular accident, and death

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Changhai Hospital, Shanghai
  - Ruijin Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - Affiliated Hospital of Jiaxing University, Zhejiang
  - Dongyang People's Hospital, Zhejiang
  - First Affiliated Hospital of Ningbo University, Zhejiang
  - Jinhua Central Hospital, Zhejiang
  - People's Hospital of Quzhou, Zhejiang
  - Shaoxing People's Hospital, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang
  - Taizhou Enze Medical Center Group, Zhejiang
  - Zhuji People's Hospital of Zhejiang Province, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided